CLINICAL TRIAL: NCT00636714
Title: Randomized Controlled Trial of Nurse-directed vs Nomogram-directed Intensive Glucose Control in the CVICU
Brief Title: Comparison of 2 Methods to Achieve Tight Glucose Control in Cardiovascular ICU Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REB 07-282c
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2017-01

CONDITIONS: Hyperglycemia in Critically Ill Patients
Keywords: intensive insulin therapy; glucose control; nurse directed; nomogram directed
MeSH Terms: interventions — Nomograms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse-directed (Experimental): Using nursing judgement to control blood glucose
  Interventions: Behavioral: Nursing judgement
- Nomogram-directed (Active Comparator): Blood glucose control directed by pre-approved paper nomogram
  Interventions: Behavioral: Nomogram

INTERVENTIONS:
Behavioral: Nursing judgement — Based on the nursing judgement, titrate insulin infusion and determine glucose check frequency to achieve a target glucose of 5-8 mmol/L
  Arms: Nurse-directed
Behavioral: Nomogram — A preprinted order outlining a nomogram with instructions for how insulin infusion should be changed based on measured glucose values and how frequent the glucose checks should be
  Arms: Nomogram-directed

SUMMARY:
There is current evidence that maintaining ICU patient's blood sugar between 4.4-6.1 saves lives. However, this is difficult to do in the ICU and carries risks of lowering the blood sugar too much. In addition, the best way to achieve this control is not known. Many strict nomograms that provide a standardized approach for nurses have been developed and validated, including one here at SMH. However, these nomograms cannot apply to all patients at all times, especially ICU patients whose needs are rapidly changing. ICU nurses are at the bedside constantly, are very familiar with their patient's needs, and have decades of experience in titrating medication doses without a nomogram to achieve a pre-determined response (i.e. medications to achieve pre-selected blood pressure). Indeed, once the bedside nurse has bought into the importance of the concept of tight glucose control and have been introduced to the nomogram here at SMH, their experience and intuition may be more adaptable to the changing needs of the patient than an inflexible paper nomogram. This study will compare glucose control using our current standard nomogram versus no nomogram (i.e. nurse directed) in order to determine whether the nomogram should continue to be used.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* adult CVICU pts
* requires insulin therapy for glucose greater than 8 mmol/L
* anticipated ICU stay > 24 hrs
* not in DKA/HHNK
* mechanically ventilated

Exclusion Criteria:

* MD refusal
* no IV access for insulin
* allergy to insulin
* DNR or moribund as determined by the clinical team

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Mean area-under-the curve for blood glucose within target per shift | over 12 hours

SECONDARY OUTCOMES:
Hypoglycemia frequency | per shift

CONTACTS AND LOCATIONS:
Overall Officials: Clarence Chant, PharmD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Chant C, Mustard M, Thorpe KE, Friedrich JO. Nurse- vs nomogram-directed glucose control in a cardiovascular intensive care unit. Am J Crit Care. 2012 Jul;21(4):270-8. doi: 10.4037/ajcc2012713. PMID 22751370